CLINICAL TRIAL: NCT05331443
Title: Effects of Ramadan Fasting on Endothelial Function
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Other Study IDs: RHIFasting
Record Dates: First submitted 2022-04-11; First posted 2022-04-15 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Fasting; Endothelial Dysfunction
Keywords: Ramadan Fasting; Endo-pat
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- participents who has the intention to fast Ramadan: subjects with at least two cardiovascular risk factors according to Framingham classification or with out any risk .
  Interventions: Diagnostic Test: Reactive hyperemia-peripheral arterial tonometry Index (RHI )

INTERVENTIONS:
Diagnostic Test: Reactive hyperemia-peripheral arterial tonometry Index (RHI ) — RHI was assessed by RH-PAT using the EndoPAT2000 system .

SUMMARY:
Include participants who intend to practice Ramadan fasting and accept to complete the three part of the study .

DETAILED DESCRIPTION:
All volunteers and stable patients that intend to fast ramadan. Each participant is examined during three separate visits.

1. The week before Ramadan (Pre-R).
2. the last week of Ramadan (R).
3. the last week of the month following Ramadan (Post-R). Participants that miss one appointement or more are exluded from the study. Patient recrutement is conducted in primary care centers of the state of Monastir, out-patients clinic (Cardiology, Endocrinology) at the emergency department of Fattouma Bourguiba university hospital after a clarified written consent.

All patients benifit of an endothelial peripheral arterial tonometry (Endo-PAT) test .

ELIGIBILITY:
Inclusion Criteria:

* Adult patient intending to fast Ramadan.

Exclusion Criteria:

* Age < 18 years old
* Hemodynamic instability.
* Myocardial infarction requiring urgent revascularization.
* Parkinsonism: tremor problem.
* Refusal, communication problem.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stable patients that intend to fast Ramadan. Each participant is examined during three planned visits. The first takes place during the month preceding Ramadan. The second during the last week of Ramadan and the third thirty days after the end of Ramadan.
  Participants that miss one appointement or more are exluded from the study. Patient recrutement is conducted in primary care centers of the state of Monastir, out-patient clinic (Cardiology, Endocrinology) at the emergency department of Fattouma Bourguiba university hospital after a clarified written consent.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in Reactive Hyperemia Index (RHI) | the day of inclusion , 10 last day of Ramadan , 1 month after Ramadan
  RHI is calculated for each participant in the day of iclusion , then it is recalculated in the two others visits.

CONTACTS AND LOCATIONS:
Overall Officials: Semir Nouira, Professor, Principal Investigator — University of Monastir
Locations (1):
- University hospital Fattouma Bourguiba, Monastir, Tunisia